CLINICAL TRIAL: NCT06528652
Title: Evaluation of Injury Profile, Core Stability and Balance in Female Hip-Hop Dancers
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Onur Yüksel ÖÇAL, Resident Physician of Sports Medicine Department, Ege University
Other Study IDs: 24-5.1T/12
Record Dates: First submitted 2024-07-17; First posted 2024-07-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Hip-Hop Dance; Athletic Injuries; Core Stability; Postural Balance
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hip-Hop (Cohort): The hip-hop dancer group will be assigned to core stability and balance performance tests as well as injury surveillance for three months.
- Non-dancer (Control): This control group will be assigned to core stability and balance performance tests only for comparison with the hip-hop dancer group and will not be subject to any injury monitoring.

SUMMARY:
The objectives of the study are to evaluate core stability and static and dynamic balance performance in adult female hip-hop dancers and compare these scores with those of healthy non-dancer females; to obtain the injury history of dancers in the last year; to follow the occurrence of new injuries for three months; and to examine the relationship between these physical performance scores and injuries.

At baseline, the hip-hop group and the non-dancer group will undergo physical performance tests.

At baseline, the hip-hop group will complete a survey asking about injury history in the past year, then complete an online survey each week for three months for injury surveillance.

DETAILED DESCRIPTION:
In dance, which is a physically demanding activity, repeated movements pose a risk of injury. Most studies investigating dance-related injuries have been conducted in the ballet discipline. The focus of this study is the hip-hop dance discipline, which has increased in popularity and has been the subject of a limited number of studies. While chronic injuries are more common in dancers, the lower extremities and low back area are most affected. Since poor core stability is noted as a risk factor for injuries in these areas, especially in females, adult female hip-hop dancers will be included in this study. Considering that balance predicts lower extremity injuries in other sports and that dancers' balance is improved with core stabilization training, balance will be evaluated in this study alongside injury surveillance and assessment of core stability. Using the survey method, the dancers' injury history within the last year will be obtained at baseline, and the injury occurrence will be followed for three months. Core stability will be assessed using McGill core endurance tests. Balance will be evaluated statically and dynamically using the unipedal stance test and the modified star excursion balance test, respectively. The relationship between core stability, balance, and injury occurrence will be examined, and furthermore, these core stability and balance results of female hip-hop dancers will be compared with the results of healthy, non-dancer females. The hip-hop dancer group will consist of hip-hop dancers registered to dance schools in İzmir. The sample size representing this group was calculated at 29. As a result of the study, the injury profile in the hip-hop dance discipline will be revealed, and it will be noticed which body parts the dancers most frequently experience problems with. It is assumed that dancers' core stability and balance results will be better than the control group, and dancers with better results will report fewer total musculoskeletal injuries at the end of a three-month follow-up. Identifying this relationship will help to make recommendations and interventions for injury prevention strategies for hip-hop dancers.

ELIGIBILITY:
Inclusion Criteria:

For the hip-hop group:

1. Being 18 years of age or older
2. Being healthy and without any initial musculoskeletal injuries
3. Competing in the adult category in the hip-hop dance discipline

For the control group:

1. Meeting the first two criteria mentioned above
2. Not being a dancer

Exclusion Criteria:

1. History of spinal or abdominal surgery
2. Pregnancy
3. Use of medications that may affect balance
4. Visual and balance impairment (for any reason)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The hip-hop dancer group will consist of adult, healthy female dancers registered to dance schools in İzmir. The control group will consist of adult, healthy, non-dancer female participants. Participants will be recruited for the study through an invitation to volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Total Number of All Physical Complaints | Upon completion of the three-month injury surveillance
  The term "injury" refers to anatomic tissue-level impairment as diagnosed by a physician that results in full-time loss from activity for one or more days beyond the day of onset. "Activity" in this definition means participation in a class, rehearsal, or performance. For those events that do not rise to the level of a reportable injury event within the surveillance system, the term "musculoskeletal complaint" should apply. However, since it was anticipated that dancers would rarely seek medical attention or continue dancing despite the problems they experienced, these two terms (injury and musculoskeletal complaints) were grouped under the title "all physical complaints."
Core Endurance Performance | At baseline
  The maximum amount of time spent maintaining the correct position in each of the flexor, extensor, and bilateral side bridge tests. The time will be recorded in seconds.
Balance Performance | At baseline
  For the assessment of static balance, the maximum amount of time and mean time spent maintaining the correct position in the unipedal stance test (performed both with eyes open and with eyes closed for both legs). The time will be recorded in seconds. Each trial will last a maximum of 45 seconds.
  For the assessment of dynamic balance, the maximum reach distance and normalized reach distance (reach divided by leg length × 100) for three directions (anterior, posterolateral, and posteromedial) in the modified star excursion balance test (for both legs). Reach distance and leg length will be measured in centimeters. A composite score is derived by averaging normalized reach distances across the three directions.

SECONDARY OUTCOMES:
Injury Occurrence Rate | Upon completion of the three-month injury surveillance
  Each participation in a class, rehearsal, or performance in which the dancer was exposed to the possibility of a dance injury constitutes one exposure. Exposure is used in the calculation of the injury rate (how often per opportunity). The number of exposures (total counts) will be recorded. The injury rate will be calculated as the total number of all physical complaints divided by the number of exposures × 1000 (e.g., 2.3 injuries per 1000 dance exposures).
  For the comparison of other studies that used dance hours in the calculation of the injury rate, total dance time will also be recorded in hours. The injury rate will also be calculated as the total number of all physical complaints divided by total dance hours × 1000 (e.g., 3.2 injuries per 1000 dance hours).
Anatomical Distribution of Injuries | Upon completion of the three-month injury surveillance
  The distribution of injuries (all physical complaints) obtained by using the marking method on the human body diagram will be expressed as a percentage of total injuries (all physical complaints) according to the body site (e.g., 30% knee, 20% low back, etc.).

OTHER OUTCOMES:
Height | At baseline
  It will be measured in centimeters with a wall-mounted stadiometer.
Weight | At baseline
  It will be measured in kilograms with a body composition analyzer.
Body Mass Index (BMI) | At baseline
  Height measurements will be converted from centimeters to meters for the calculation. BMI will be calculated as weight (in kilograms) / height (in meters) x height (in meters).
Body Fat (BF) | At baseline
  It will be measured with a body composition analyzer and shown as a percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Onur Y ÖÇAL, Resident, Principal Investigator — Ege University Faculty of Medicine, Department of Sports Medicine; Cengizhan ÖZGÜRBÜZ, Professor, Study Chair — Ege University Faculty of Medicine, Department of Sports Medicine
Locations (1):
- Ege University Faculty of Medicine, Department of Sports Medicine, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambegaonkar JP, Hansen-Honeycutt J, Wiese KR, Cavanagh CM, Caswell SV, Ambegaonkar SJ, Martin J. Female Collegiate Dancers' Physical Fitness across Their Four-Year Programs: A Prospective Analysis. J Funct Morphol Kinesiol. 2023 Jul 17;8(3):98. doi: 10.3390/jfmk8030098. PMID 37489311
- [Background] Ursej E, Zaletel P. Injury Occurrence in Modern and Hip-Hop Dancers: A Systematic Literature Review. Zdr Varst. 2020 Jun 25;59(3):195-201. doi: 10.2478/sjph-2020-0025. eCollection 2020 Sep. PMID 32952721
- [Background] Jubb C, Bell L, Cimelli S, Wolman R. Injury Patterns in Hip Hop Dancers. J Dance Med Sci. 2019 Dec 15;23(4):145-149. doi: 10.12678/1089-313X.23.4.145. PMID 31775952
- [Background] Ursej E, Sekulic D, Prus D, Gabrilo G, Zaletel P. Investigating the Prevalence and Predictors of Injury Occurrence in Competitive Hip Hop Dancers: Prospective Analysis. Int J Environ Res Public Health. 2019 Sep 3;16(17):3214. doi: 10.3390/ijerph16173214. PMID 31484349
- [Background] Ojofeitimi S, Bronner S, Woo H. Injury incidence in hip hop dance. Scand J Med Sci Sports. 2012 Jun;22(3):347-55. doi: 10.1111/j.1600-0838.2010.01173.x. Epub 2010 Aug 30. PMID 20807386
- [Background] Tjukov O, Engeroff T, Vogt L, Banzer W, Niederer D. Injury Profile of Hip-Hop Dancers. J Dance Med Sci. 2020 Jun 15;24(2):66-72. doi: 10.12678/1089-313X.24.2.66. PMID 32456761
- [Background] Dang Y, Chen R, Koutedakis Y, Wyon MA. The Efficacy of Physical Fitness Training on Dance Injury: A Systematic Review. Int J Sports Med. 2023 Feb;44(2):108-116. doi: 10.1055/a-1930-5376. Epub 2022 Aug 24. PMID 36002027
- [Background] Rickman AM, Ambegaonkar JP, Cortes N. Core stability: implications for dance injuries. Med Probl Perform Art. 2012 Sep;27(3):159-64. PMID 22983134
- [Background] Huxel Bliven KC, Anderson BE. Core stability training for injury prevention. Sports Health. 2013 Nov;5(6):514-22. doi: 10.1177/1941738113481200. PMID 24427426
- [Background] Russell JA. Preventing dance injuries: current perspectives. Open Access J Sports Med. 2013 Sep 30;4:199-210. doi: 10.2147/OAJSM.S36529. PMID 24379726
- [Background] Chatfield SJ, Krasnow DH, Herman A, Blessing G. A Descriptive Analysis of Kinematic and Electromyographic Relationships of the Core during Forward Stepping in Beginning and Expert Dancers. Journal of Dance Medicine & Science. 2007;11(3):76-84. doi:10.1177/1089313X0701100303
- [Background] Watson T, Graning J, McPherson S, Carter E, Edwards J, Melcher I, Burgess T. DANCE, BALANCE AND CORE MUSCLE PERFORMANCE MEASURES ARE IMPROVED FOLLOWING A 9-WEEK CORE STABILIZATION TRAINING PROGRAM AMONG COMPETITIVE COLLEGIATE Dancers. Int J Sports Phys Ther. 2017 Feb;12(1):25-41. PMID 28217414
- [Background] Li L, Waldhelm A. Endurance tests are the most reliable core stability related measurements. J Sport Health Sci. 2012; 1:121-8. doi: 10.1016/j.jshs.2012.07.007.
- [Background] McGill SM, Childs A, Liebenson C. Endurance times for low back stabilization exercises: clinical targets for testing and training from a normal database. Arch Phys Med Rehabil. 1999 Aug;80(8):941-4. doi: 10.1016/s0003-9993(99)90087-4. PMID 10453772
- [Background] del Pozo-Cruz B, Mocholi MH, del Pozo-Cruz J, Parraca JA, Adsuar JC, Gusi N. Reliability and validity of lumbar and abdominal trunk muscle endurance tests in office workers with nonspecific subacute low back pain. J Back Musculoskelet Rehabil. 2014;27(4):399-408. doi: 10.3233/BMR-140460. PMID 24561788
- [Background] Swain C, Redding E. Trunk muscle endurance and low back pain in female dance students. J Dance Med Sci. 2014;18(2):62-6. doi: 10.12678/1089-313X.18.2.62. PMID 24844422
- [Background] Ambegaonkar JP, Mettinger LM, Caswell SV, Burtt A, Cortes N. Relationships between core endurance, hip strength, and balance in collegiate female athletes. Int J Sports Phys Ther. 2014 Oct;9(5):604-16. PMID 25328823
- [Background] Latimer J, Maher CG, Refshauge K, Colaco I. The reliability and validity of the Biering-Sorensen test in asymptomatic subjects and subjects reporting current or previous nonspecific low back pain. Spine (Phila Pa 1976). 1999 Oct 15;24(20):2085-9; discussion 2090. doi: 10.1097/00007632-199910150-00004. PMID 10543003
- [Background] Paris-Alemany A, Torres-Palomino A, Marino L, Calvo-Lobo C, Gadea-Mateos L, La Touche R. Comparison of lumbopelvic and dynamic stability between dancers and non-dancers. Phys Ther Sport. 2018 Sep;33:33-39. doi: 10.1016/j.ptsp.2018.06.010. Epub 2018 Jul 2. PMID 29982036
- [Background] Plisky PJ, Gorman PP, Butler RJ, Kiesel KB, Underwood FB, Elkins B. The reliability of an instrumented device for measuring components of the star excursion balance test. N Am J Sports Phys Ther. 2009 May;4(2):92-9. PMID 21509114
- [Background] Gribble, P. A., & Hertel, J. (2003). Considerations for Normalizing Measures of the Star Excursion Balance Test. Measurement in Physical Education and Exercise Science, 7(2), 89-100. https://doi.org/10.1207/S15327841MPEE0702_3
- [Background] Plisky PJ, Rauh MJ, Kaminski TW, Underwood FB. Star Excursion Balance Test as a predictor of lower extremity injury in high school basketball players. J Orthop Sports Phys Ther. 2006 Dec;36(12):911-9. doi: 10.2519/jospt.2006.2244. PMID 17193868
- [Background] Smith CA, Chimera NJ, Warren M. Association of y balance test reach asymmetry and injury in division I athletes. Med Sci Sports Exerc. 2015 Jan;47(1):136-41. doi: 10.1249/MSS.0000000000000380. PMID 24870573
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Liederbach M, Hagins M, Gamboa JM, Welsh TM. Assessing and Reporting Dancer Capacities, Risk Factors, and Injuries: Recommendations from the IADMS Standard Measures Consensus Initiative. J Dance Med Sci. 2012 Dec;16(4):139-53. PMID 26731091